CLINICAL TRIAL: NCT01240382
Title: Double-masked Comparison Study of DE-089 Ophthalmic Solution in Patients With Dry Eye (Multi-center Study, in Comparison to 0.1% Sodium Hyaluronate Ophthalmic Solution) - Phase III Confirmatory Study -
Brief Title: Phase III Confirmatory Study of DE-089 Ophthalmic Solution in Patients With Dry Eye
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Santen Pharmaceutical Co., Ltd. (Industry)
Other Study IDs: 00890602
Record Dates: First submitted 2010-11-12; First posted 2010-11-15 (Estimated); Results first posted 2014-08-08 (Estimated); Last update posted 2014-08-13 (Estimated); Status verified 2014-08

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

ARMS (2):
- 3% DE-089 (Experimental)
  Interventions: Drug: 3% DE-089 ophthalmic solution
- 0.1% HA (Active Comparator)
  Interventions: Drug: 0.1% sodium hyaluronate ophthalmic solution

INTERVENTIONS:
Drug: 3% DE-089 ophthalmic solution
  Arms: 3% DE-089
Drug: 0.1% sodium hyaluronate ophthalmic solution
  Arms: 0.1% HA

SUMMARY:
To investigate that the efficacy of 3% DE-089 ophthalmic solution (one drop at a time, 6 times daily, 4 weeks topical administration), in comparison to 0.1% sodium hyaluronate ophthalmic solution (0.1% HA) (one drop at a time, 6 times daily, 4 weeks topical administration), is at least non-inferior in the change in fluorescein staining score, and is superior in the change in Rose bengal score, in a multicenter, double-masked, parallel-group comparison study. Safety profile will likewise be compared.

ELIGIBILITY:
Inclusion Criteria:

* Those who show:

  * Keratoconjunctival disorder confirmed with vital dye staining
  * Abnormal Schirmer score results

Exclusion Criteria:

* Eye disease that needs therapy other than that for dry eye
* Those who need to wear contact lenses during the clinical study

Min Age: 20 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 332 (Actual)
Dates: Primary Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Santen study sites, Osaka, Osaka, Japan

REFERENCES:
- [Derived] Takamura E, Tsubota K, Watanabe H, Ohashi Y; Diquafosol Ophthalmic Solution Phase 3 Study Group. A randomised, double-masked comparison study of diquafosol versus sodium hyaluronate ophthalmic solutions in dry eye patients. Br J Ophthalmol. 2012 Oct;96(10):1310-5. doi: 10.1136/bjophthalmol-2011-301448. Epub 2012 Aug 21. PMID 22914501

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Informed consent was obtained from 332 patients, of whom 287 were randomized and prescribed the study drug.
Groups:
- 3% DE-089: 3% DE-089 ophthalmic solution
- 0.1% HA: 0.1% sodium hyaluronate ophthalmic solution
Period: Overall Study
Arm/Group | 3% DE-089 | 0.1% HA
Started | 144 | 143
Completed | 142 | 139
Not Completed | 2 | 4
Not completed — Adverse Event | 2 | 1
Not completed — Lack of Efficacy | 0 | 2
Not completed — Fear of adverse events | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 3% DE-089 | 0.1% HA | Total
Number analyzed (Participants) | 144 | 143 | 287
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.3 (17.1) | 57.0 (16.8) | 56.1 (16.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 120 | 125 | 245
  Male | 24 | 18 | 42

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Fluorescein Staining Score From Baseline
Description: Fluorescein staining was scored according to the protocol by Shimmura et al. The cornea was divided into 3 equal zones: upper, middle, and lower. Each zone had a staining score ranging between 0 and 3 points, with minimum and maximum total staining scores ranging between 0 and 9 points. 0 is better.
  The degree of staining with Fluorescein dyes was scored as follows: 0 = no staining, 1= staining of less than half of the area, 2= staining of more than half of the area, 3= staining in the whole area.
Time Frame: Baseline and 4-week (discontinued (LOCF))
Population: Efficacy analysis was performed full analysis set (FAS). In 0.1% sodium hyaluronate ophthalmic solution group, 1 subject was excluded from analysis because there was no available efficacy data in fluorescein staining.
Measure: Mean (Standard Deviation); unit: points
Arm/Group | 3% DE-089 | 0.1% HA
Number analyzed (Participants) | 144 | 142
points | -2.12 (1.66) | -2.08 (1.52)
Statistical Analysis 1: Comparison: 3% DE-089 vs 0.1% HA; Test type: Non-Inferiority or Equivalence — Non-inferiority in mean change in fluorescein staining score from baseline was assessed on the non-inferiority margin (0.34) with the upper limit of the confidence interval of the difference between the 2 treatment groups; l; Median Difference (Final Values) = -0.03, 95% CI [-0.405 to 0.338]

2. Primary Outcome: Mean Change in Rose Bengal Staining Score From Baseline
Description: Rose bengal staining were scored according to the protocol by Shimmura et al. The ocular surface was divided into 5 zones: nasal and temporal conjunctival, and upper, middle, and lower corneal areas. A staining score between 0 and 3 points was used in each zone, with the minimum and maximum total staining scores ranging between 0 and 15 points.0 is better.
  The degree of staining with Rose bengal dyes was scored as follows: 0 = no staining, 1= staining of less than half of the area, 2= staining of more than half of the area, 3= staining in the whole area.
Time Frame: Baseline and 4-week (discontinued (LOCF))
Population: Efficacy analysis was performed full analysis set (FAS). In 0.1% sodium hyaluronate ophthalmic solution group, 2 subjects were excluded from analysis because there was no available efficacy data in rose bengal staining.
Measure: Mean (Standard Deviation); unit: points
Arm/Group | 3% DE-089 | 0.1% HA
Number analyzed (Participants) | 144 | 141
points | -3.06 (2.27) | -2.38 (2.08)
Statistical Analysis 1: Comparison: 3% DE-089 vs 0.1% HA; Test type: Superiority or Other; p = 0.010, t-test, 2 sided; Median Difference (Final Values) = -0.67, 95% CI [-1.18 to -0.67]

ADVERSE EVENTS:
Arm/Group | 3% DE-089 | 0.1% HA
Serious Adverse Events (participants affected / at risk) | 0/144 | 1/143
Other Adverse Events (participants affected / at risk) | 9/144 | 1/143
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 3% DE-089 (N=144) | 0.1% HA (N=143)
Gastrointestinal bleeding (Gastrointestinal disorders) | 0 | 1 — There was a serious adverse event in 0.1% sodium hyaluronate ophthalmic solution group
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 3% DE-089 (N=144) | 0.1% HA (N=143)
Eye irritation (Eye disorders) | 9 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No